CLINICAL TRIAL: NCT02188914
Title: Neurobiología Del Consumo de Substancias Psicoactivas: PET-CT- Inhalables
Brief Title: Brain Imaging Studies of the Effect of Inhalant Use Disorder
Status: Completed | Type: Observational
Sponsor: Miguel Ángel Mendoza Meléndez (Other Government)
Collaborators: National Institute of Neurology and Neurosurgery, Mexico (Other)
Responsible Party: Sponsor-Investigator, Miguel Ángel Mendoza Meléndez, Director of Research and Evaluation, Instituto para la Atención y Prevención de las Adicciones en la Ciudad de México
Organization: Instituto para la Atención y Prevención de las Adicciones en la Ciudad de México (Other Government)
Other Study IDs: 11/13 protocol
Record Dates: First submitted 2014-07-09; First posted 2014-07-14 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Inhalant Use Disorder
Keywords: Inhalant use disorder; Positron emission tomography; Magnetic Resonance Imaging; Executive functions assessment; Transcriptome
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — cDNA obtained from reversal transcription of RNA isolated from periferical blood cells
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Inhalant use disorder group: Subjects must have a diagnosis of inhalant use disorder, according to the DSM-5, who are under a treatment program for addictive disorders.
  Interventions: Radiation: Positron emission tomography scan; Other: Magnetic resonance imaging
- Normal control group: Normal control without a history of drug abuse or dependency.
  Interventions: Radiation: Positron emission tomography scan; Other: Magnetic resonance imaging

INTERVENTIONS:
Radiation: Positron emission tomography scan
Other: Magnetic resonance imaging

SUMMARY:
Inhalants substance misuse is an important public health problem whose prevalence is approximately 1% in the general population and 7% among high school students in Mexico. Furthermore Inhalants substance misuse has increased in the recent years (Villatoro et al., 2011). According to the Diagnostic and Statistical Manual of Mental Disorders fifth edition (DSM-5) inhalant use disorder is a problematic pattern of use of a hydrocarbon-based inhalant substance leading to clinically significant impairment or distress. There are studies to suggest that long-term exposure to inhalants is associated with structural brain abnormalities, as well as neuropsychological impairments. However many of these studies have been limited to the gross anatomical report, therefore is necessary the use of complimentary techniques which provide a better understanding of brain. To the date there is no evidence of the use of positron emission tomography, and there are few studies have employed other magnetic resonance imaging methodologies such as diffusion tensor imaging that can be used to know the metabolic activity and white matter tract integrity respectively in inhalant use disorder participants. The purpose of this study is evaluates the effects of the inhalant use disorder in the brain. The investigators will be using positron emission tomography (PET), Magnetic Resonance Imaging (MRI) and diffusion tensor imaging (DTI). As well as, this study will examine the impact of inhalants consumption on executive function performance and the transcriptomic changes associated with inhalants consumption. The investigators hope that the data gathered from this study will lead to the development of more effective treatments

ELIGIBILITY:
Inclusion Criteria:

* Males between 18 to 40 years old.
* Subjects must have a diagnosis of inhalant use disorder who are under a treatment program for addictive disorders or normal control without a history of drug abuse or dependency. Control participants must be matches with the inhalant use disorder participants according to age and years of education.
* Subjects in both the inhalant use disorder and control groups will be volunteers who signed informed consent.

Exclusion Criteria:

* Epilepsy or clinically relevant seizures in the last year
* Cognitive impairment evaluated through Mini-Mental State Examination
* Psychosis
* Manic or hypomanic episode
* Moderate or severe suicide risk
* Panic disorder
* Claustrophobia: Subjects will be questioned about their potential discomfort in being in an enclosed space, such as a PET or MRI scanner.
* History of head trauma with loss of consciousness > 30 min.
* Neurological surgical procedures
* Diabetes
* Positive test for hippuric acid
* Current use of antipsychotic medication
* Current illnesses, painful conditions or other disorders, which in the judgment of the investigators, might invalidate the scientific goals of the study or pose undesirable difficulties or risks for subjects
* In the case for magnetic resonance imaging, Individuals who would be unable to undergo a MRI scan, for example, individuals who have metal clips in their body, metallic prostheses (i.e., replacement body parts, such as a hip joint), a pacemaker, or other pieces of metal in their body (shrapnel, metal filings, etc.).

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants in inhalant use disorder treatment program or Normal Control Subjects volunteers
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2016-07-30 (Actual); Study Completion 2016-07-30 (Actual)

PRIMARY OUTCOMES:
Brain metabolic activity | Baseline
  Determine if the inhalant use disorder participants have different brain metabolic activity than healthy controls
Abnormalities in the fractional anisotropy | Baseline
  Determine if the inhalant use disorder participants show abnormalities in the fractional anisotropy than healthy controls
Behavioral performance measures on the executive functions | Baseline
  Determine if the inhalant use disorder participants show neuropsychological impairments relative to healthy controls in attention and executive functions
Severity inhalant use disorder | Baseline
  Determine if the brain metabolic activity is associated with the severity inhalant use disorder.
  Determine if the abnormalities in the fractional anisotropy are associated with the severity inhalant use disorder.
Ratings and scores in the Pittsburgh Sleep Quality Index | Baseline
  The proportion of participants that have good or bad sleep Quality.
Age at which inhalants use began | Baseline
  Determine if the brain metabolic activity is associated with the age at which inhalants use began.
  Determine if the abnormalities in the fractional anisotropy are associated with the age at which inhalants use began.
Duration of regular inhalant use | Baseline
  Determine if the brain metabolic activity is associated with the duration of regular inhalant use.
  Determine if the abnormalities in the fractional anisotropy are associated with the duration of regular inhalant use.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Ángel Mendoza Meléndez, MD, MPH, Principal Investigator — Institute for Attention and Prevention of Addictions in Mexico City; Nora Estela Kerik Rotenberg, MD, Principal Investigator — National Institute of Neurology and Neurosurgery Manuel Velasco Suárez.
Locations (1):
- National Institute of Neurology and Neurosurgery Manuel Velasco Suarez, Mexico City, Mexico

REFERENCES:
- [Background] Villatoro JA, Cruz SL, Ortiz A, Medina-Mora ME. Volatile substance misuse in Mexico: correlates and trends. Subst Use Misuse. 2011;46 Suppl 1:40-5. doi: 10.3109/10826084.2011.580205. PMID 21609144
- [Background] Yucel M, Takagi M, Walterfang M, Lubman DI. Toluene misuse and long-term harms: a systematic review of the neuropsychological and neuroimaging literature. Neurosci Biobehav Rev. 2008 Jul;32(5):910-26. doi: 10.1016/j.neubiorev.2008.01.006. Epub 2008 Mar 27. PMID 18456329
- [Background] Aydin K, Sencer S, Demir T, Ogel K, Tunaci A, Minareci O. Cranial MR findings in chronic toluene abuse by inhalation. AJNR Am J Neuroradiol. 2002 Aug;23(7):1173-9. PMID 12169477
- [Background] Brouette T, Anton R. Clinical review of inhalants. Am J Addict. 2001 Winter;10(1):79-94. doi: 10.1080/105504901750160529. PMID 11268830
- [Background] Takagi M, Lubman DI, Walterfang M, Barton S, Reutens D, Wood A, Yucel M. Corpus callosum size and shape alterations in adolescent inhalant users. Addict Biol. 2013 Sep;18(5):851-4. doi: 10.1111/j.1369-1600.2011.00364.x. Epub 2011 Sep 29. PMID 21955104
- [Background] Yucel M, Zalesky A, Takagi MJ, Bora E, Fornito A, Ditchfield M, Egan GF, Pantelis C, Lubman DI. White-matter abnormalities in adolescents with long-term inhalant and cannabis use: a diffusion magnetic resonance imaging study. J Psychiatry Neurosci. 2010 Nov;35(6):409-12. doi: 10.1503/jpn.090177. PMID 20731960
- [Background] Volkow ND, Fowler JS, Wang GJ. Positron emission tomography and single-photon emission computed tomography in substance abuse research. Semin Nucl Med. 2003 Apr;33(2):114-28. doi: 10.1053/snuc.2003.127300. PMID 12756644